CLINICAL TRIAL: NCT03013569
Title: Can Spontaneous Fetal EEG Be Recorded During Labor Using the Established Fetal Scalp Electrode Heart Rate Monitoring System?
Brief Title: Spontaneous Fetal EEG Recording During Labor
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Martin Frasch, Research Assistant Professor, Obstetrics and Gynecology, University of Washington
Other Study IDs: STUDY00003276
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Abnormal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot feasibility study for a new application of an approved fetal heart rate monitoring device system. The objective of this study is to validate the feasibility of acquiring the new modality of human fetal bioelectrical activity, EEG, derived from the routinely used scalp fetal heart rate (FHR) monitor.

DETAILED DESCRIPTION:
The investigators' objective is to validate the feasibility of acquiring the new modality of human fetal bioelectrical activity, EEG, derived from the routinely used scalp FHR monitor.

The investigators expect that in some newborns acidemia will be detected based on cord blood pH. In these babies, the investigators will trace back the EEG recordings to further validate whether the EEG - FHR patterns were predictive of this outcome. In fetal sheep model of human labour the investigators were able to see the onset of acidemia <55 min ahead of severe drop of pH to <7.00. This corresponded to an average pH of 7.20.

The investigators hypothesize that they will be able to acquire fetal EEG during labour such that the normal behavioural sleep states will be observed and their disruption, followed by emergence of the pathognomonic EEG-FHR pattern will be seen with incipient acidemia.

At-risk pregnant women routinely admitted for intrapartum monitoring will be asked to consent when the Fetal Scalp Monitor (FSM) is placed. The attachment will be such that no direct contact to mother or baby will be established and hence no current from device to the mother or the baby will be possible. The EEG fetal health monitoring device is attached to the routinely used fetal heart rate (FHR) GE HC Corometrix 250cx monitor. The EEG recording will commence only once the FSM is attached; the attachment of the FSM will be performed based on medical necessity, not based on the need to record EEG.

Duration of recording will be dependent on the labour duration. However, the investigators will seek for a minimum of 30 minutes and continue as long as medically possible per subject.

Fetal EEG will be analyzed as published. The quickest reference to the analytical approach is given here: http://dx.doi.org/10.1371/journal.pone.0108119.g001

Cord blood gas at delivery will be recorded from electronic medical record, as it is taken routinely at birth. Basic maternal and neonatal clinical characteristics (BMI, APGAR scores, number of pregnancies and live births, maternal and fetal ages at birth), will also be taken from the medical record.

b. Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you or your team have that supports the feasibility and/or safety of this study. Nine years of research and development to show that fetal EEG measurements can predict the level of acidemia at birth. Safety testing performed on site successfully for recording fetal EEG during labor as described.

ELIGIBILITY:
Inclusion Criteria:

Women in labor, with medical complications of pregnancy, such as IUGR, hypertension, diabetes, or obesity (BMI over 30).

Exclusion Criteria:

1. Maternal or fetal infection or bleeding disorder;
2. Birth through Caesarian section will only be excluded if decided a priori;
3. Non-English speaking.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women of reproductive age in labor at term
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-01; Primary Completion 2022-12 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Recording spontaneous EEG during labor | 12 month recruitment period
  The investigators will record spontaneous fetal EEG activity during labor using a custom-build IRB-approved fetal EEG device. The validity of the recorded data will be analyzed based on the physiological characteristics of the data such as amplitude and frequency properties as well as the behavioral state architecture (duration of low voltage/high frequency and high voltage/low frequency states as well as of the indeterminate states). The data will be analyzed in conjunction with the accompanying fetal heart rate recordings which also show behavioral state fluctuations.

SECONDARY OUTCOMES:
Fetal acidemia | 12 month recruitment period
  EEG recordings will be used to validate whether the EEG-FHR patterns are predictive of fetal acidemia intrapartum

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Frasch, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, Durosier LD, Ross MG, Richardson BS, Frasch MG. Online detection of fetal acidemia during labour by testing synchronization of EEG and heart rate: a prospective study in fetal sheep. PLoS One. 2014 Sep 30;9(9):e108119. doi: 10.1371/journal.pone.0108119. eCollection 2014. PMID 25268842
- [Background] Frasch MG, Durosier LD, Gold N, Cao M, Matushewski B, Keenliside L, Louzoun Y, Ross MG, Richardson BS. Adaptive shut-down of EEG activity predicts critical acidemia in the near-term ovine fetus. Physiol Rep. 2015 Jul;3(7):e12435. doi: 10.14814/phy2.12435. PMID 26149280
- [Background] Xu A, Durosier LD, Ross MG, Hammond R, Richardson BS, Frasch MG. Adaptive brain shut-down counteracts neuroinflammation in the near-term ovine fetus. Front Neurol. 2014 Jun 30;5:110. doi: 10.3389/fneur.2014.00110. eCollection 2014. PMID 25071698
- [Background] Frasch MG, Keen AE, Gagnon R, Ross MG, Richardson BS. Monitoring fetal electrocortical activity during labour for predicting worsening acidemia: a prospective study in the ovine fetus near term. PLoS One. 2011;6(7):e22100. doi: 10.1371/journal.pone.0022100. Epub 2011 Jul 15. PMID 21789218
- [Result] Castel A, Frank YS, Feltner J, Karp FB, Albright CM, Frasch MG. Monitoring Fetal Electroencephalogram Intrapartum: A Systematic Literature Review. Front Pediatr. 2020 Sep 11;8:584. doi: 10.3389/fped.2020.00584. eCollection 2020. PMID 33042922
- See also: The website of the laboratory of Dr. Frasch, the PI on the study — https://FraschLab.org